CLINICAL TRIAL: NCT00862836
Title: Addition of Vandetanib to Standard Therapy (Pegliposomal Doxorubicin) in Patients With Recurrent Ovarian Cancer. A Multicentre Phase I / Randomized Phase II Study
Brief Title: Addition of Vandetanib to Standard Therapy Pegliposomal Doxorubicin (PLD)
Acronym: ZACFAST
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00083; 2008-005557-38 (EudraCT Number)
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Ovarian Cancer
Keywords: ZD6474; Vandetanib; Zactima; Ovarian Cancer; Phase I; Phase II; Randomized; Safety
MeSH Terms: conditions — Ovarian Neoplasms | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vandetanib added to standard therapy (pegliposomal doxorubicin)
  Interventions: Drug: Vandetanib

INTERVENTIONS:
Drug: Vandetanib — 100mg doses orally, once daily
  Other Names: Zactima

SUMMARY:
This multi-centre, non-randomized open phase I/randomized phase II study will be conducted in 70 patients (10 in phase I, 60 in phase II) with platinum-refractory recurrent epithelial cancer of the ovary, fallopian tube or peritoneum. A total of approximately 5 national centers will participate in phase I of the study. If the starting criteria for phase II of the study are met at the end of phase I, a total of approximately 20 national centers will participate in phase II of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically documented invasive epithelial ovarian carcinoma, cancer of the fallopian tube or the peritoneum refractory to platinum-based chemotherapy or with partially platinum sensitive disease.
* Planned therapy with pegylated liposomal doxorubicin 50 mg/m² for recurrent platinum-refractory ovarian cancer.
* Patients with a progression-free-interval of 6 to 12 months after platinum-based chemotherapy are only eligible if a further course of platinum-based combination chemotherapy is not possible as judged by the investigator(s).
* Patients must have received at least one previous platinum- and taxane-based chemotherapy regimen.

Exclusion Criteria:

* Brain metastases or spinal cord compression, unless treated at least 4 weeks before first dose and stable without steroid treatment for 10 days
* Any concomitant medications that may cause QTc prolongation or induce Torsades de Pointes or induce CYP3A4 function
* Treatment with mouse-antibodies in patients with evaluable disease and CA-125 progressive disease in the last 3 months. These patients are only eligible in case of measurable disease according to RECIST or cytological/histological proven relapse
* More than two prior lines of chemotherapy.
* Any chemotherapy or other systemic anti-cancer therapy within four weeks prior to randomization.
* Radiation therapy within the last 4 weeks prior to randomization (with the exception of palliative radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- Germany (5):
  - Research Site, Ulm, Baden-Wurttemberg
  - Research Site, Wiesbaden, Hesse
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Kiel, Schleswig-Holstein
  - Research Site, Berlin

REFERENCES:
- [Derived] Harter P, Sehouli J, Kimmig R, Rau J, Hilpert F, Kurzeder C, Elser G, du Bois A. Addition of vandetanib to pegylated liposomal doxorubicin (PLD) in patients with recurrent ovarian cancer. A randomized phase I/II study of the AGO Study Group (AGO-OVAR 2.13). Invest New Drugs. 2013 Dec;31(6):1499-504. doi: 10.1007/s10637-013-0011-3. Epub 2013 Sep 5. PMID 24005613

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I of the trial consisted of a safety run-in phase of 10 patients with histologically confirmed, epithelial ovarian carcinoma, cancer of the fallopian tube or the peritoneum refractory or partially sensitive to platinum-based therapy evaluable for at least 2 cycles.
  Phase II of the trial was not conducted.
Groups:
- Vandetanib 100 mg: Once daily oral Vandetanib 100 mg added to standard therapy (pegylated liposomal doxorubicin 50 mg/m2 iv every 4 weeks)
Period: Overall Study
Arm/Group | Vandetanib 100 mg
Started | 15
Evaluable for Safety/Toxicity | 14 (1 patient withdrew consent before first cycle)
Evaluable for Activity (Tumour Response) | 10
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vandetanib 100 mg
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Description (on the Basis of the Safety Set): Safety and Tolerability by Means of the Incidence and Type of Adverse Events (AEs).
Description: Number of participants with at least 1 adverse event of grade 3 or higher (CTCAE grade 3=severe, CTCAE grade 4=life threatening/disabling, CTCAE grade 5=death, as defined by National Cancer Institute CTCAE, Version 3)
Time Frame: From date of registration (Informed Consent Form completed) to date of last vist, up to 18 months.
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg
Number analyzed (Participants) | 14
Participants | 9

2. Secondary Outcome: Evaluation (for ITT Set): Clinical Activity of Once Daily Oral Vandetanib 100 mg When Added to Standard Therapy (See Above), by Assessment of Progression Free Survival (PFS).
Description: Progression Free Survival: Progression is defined using RECIST, as a measurable increase of at least 20% in the sum of longest diameters of target lesions or unequivocal progression of non-target lesions, or the appearance of new lesions, since baseline.
Time Frame: From date of registration (Informed Consent Form completed) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 100 mg
Number analyzed (Participants) | 10
Months | 6.7 [0.87 to 13.73]

3. Secondary Outcome: Evaluation (for ITT Set): Clinical Activity of Once Daily Oral Vandetanib 100 mg When Added to Standard Therapy (See Above), by Assessment of Overall Survival (OS).
Description: Median overall survival (OS)
Time Frame: From date of registration (Informed Consent Form completed) until the date of death.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib 100 mg
Number analyzed (Participants) | 10
Months | 11.1 [2.17 to 14.93]

4. Primary Outcome: Description (on the Basis of the Safety Set): Safety and Tolerability by Means of Clinically Significant Laboratory Abnormalities.
Description: Number of patients with elevated liver enzymes grade 3 (CTCAE grade 3=severe, CTCAE grade 4=life threatening).
Time Frame: From date of registration (Informed Consent Form completed) to date of last vist, up to 18 months.
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg
Number analyzed (Participants) | 14
Participants | 3

5. Primary Outcome: Description (on the Basis of the Safety Set): Safety and Tolerability by Means of the Incidence and Type of Adverse Events (AEs). Number of Participants With Dermatologic Skin Reactions Grade 3/4.
Description: Number of participants with dermatologic skin reactions grade 3/4 (CTCAE grade 3= severe, CTCAE grade 4=life threatening)
Time Frame: From date of registration (Informed Consent Form completed) to date of last vist, up to 18 months.
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg
Number analyzed (Participants) | 14
Participants | 5

6. Primary Outcome: Description (on the Basis of the Safety Set): Safety and Tolerability by Means of the Incidence and Type of Adverse Events (AEs). Number of Participants With Palmar-plantar Erythrodysesthesia (PPE) Grade 3/4.
Description: Number of participants with palmar-plantar erythrodysesthesia (PPE) grade 3/4 (CTCAE grade 3=severe skin changes with pain, CTCAE grade 4=life threatening).
Time Frame: From date of registration (Informed Consent Form completed) to date of last vist, up to 18 months.
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg
Number analyzed (Participants) | 14
Participants | 5

7. Primary Outcome: Description (on the Basis of the Safety Set): Safety and Tolerability by Means of the Incidence and Type of Adverse Events (AEs). Number of Participants With Mucositis Grade 3.
Description: Number of participants with mucositis grade 3 (CTCAE grade 3=severe pain interfering with oral intake)
Time Frame: From date of registration (Informed Consent Form completed) to date of last vist, up to 18 months.
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg
Number analyzed (Participants) | 14
Participants | 2

8. Primary Outcome: Description (on the Basis of the Safety Set): Safety and Tolerability by Means of Clinically Significant Laboratory Abnormalities. Number of Participants With Neutropenia Grade 3/4.
Description: Number of participants with neutropenia grade 3/4 (CTCAE grade 3=severe, CTCAE grade 4=life threatening).
Time Frame: From date of registration (Informed Consent Form completed) to date of last vist, up to 18 months.
Measure: Number; unit: Participants
Arm/Group | Vandetanib 100 mg
Number analyzed (Participants) | 14
Participants | 2

ADVERSE EVENTS:
Arm/Group | Vandetanib 100 mg
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib 100 mg (N=14)
Arrhythmia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib 100 mg (N=14)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Oesophagitis (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Oesophageal pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Mucosal inflammation (General disorders) | 6
Chills (General disorders) | 1
Mucosal dryness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Gamma-glutamyltransferase (Investigations) | 6
Rhinitis (Infections and infestations) | 1
Aspartate aminotransferase (Investigations) | 5
White blood cell count (Investigations) | 5
Alanine aminotransferase (Investigations) | 4
Blood alkaline phosphatase (Investigations) | 4
Blood creatinine (Investigations) | 3
Blood lactate dehydrogenase (Investigations) | 3
Haemoglobin (Investigations) | 3
Blood glucose (Investigations) | 2
Monocyte count (Investigations) | 2
Protein total (Investigations) | 2
Activated partial thromboplastin time (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin (Investigations) | 1
Blood calcium (Investigations) | 1
Blood chloride (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood magnesium decreased (Investigations) | 1
Blood potassium (Investigations) | 1
Haematocrit (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Monocyte count decreased (Investigations) | 1
Neutrophil count (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Prothrombin time (Investigations) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Peripheral sensory neuropath (Nervous system disorders) | 1
Sleep disorder (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Chromaturia (Psychiatric disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
International normalised ratio (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.